CLINICAL TRIAL: NCT06980558
Title: Effect of Progressive Relaxation Exercises on Sleep Quality in Patients Undergoing Urological Surgery
Brief Title: Effect of Progressive Muscle Exercises on Sleep in Urological Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Cagla Toprak, Dr, Atlas University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05/01
Record Dates: First submitted 2025-05-04; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Surgery; Sleep Quality; Sleep
Keywords: urological Surgery; sleep quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): The individual will be given a position where communication can be easily established and where he/she feels comfortable. The content of the progressive relaxation exercise (PGE) will be explained to the patient. The 30-minute PGE application will be provided with verbal warnings.
  Interventions: Other: Progressive relaxation exercises
- Control group (No Intervention): Patients will receive routine nursing care in the ward.

INTERVENTIONS:
Other: Progressive relaxation exercises — Sit or lie down comfortably and close your eyes.
  * Feel the rhythm of your breathing.
  * Breathe in through your nose and out through your mouth throughout the process.
  * Relax as much as you can.
  * Get rid of negative thoughts in your mind.
  * Stretch your hands by hanging your arms down to your sides, tighten your fists as much as you can and then open them and let them relax.
  Arms: Exercise group

SUMMARY:
Patients undergoing urological surgery are usually elderly individuals and may experience sleep problems due to factors such as fear of death, anesthesia, and uncertainty. Insomnia can also cause problems such as delayed wound healing, increased pain, tension, and difficulty complying with treatment. This study aimed to improve sleep quality by performing gradual muscle exercises on patients undergoing urological surgery.

DETAILED DESCRIPTION:
Urological surgery is a type of surgery that is usually performed on elderly individuals and can cause serious sleep problems in the pre- and post-operative period. While these patients experience sleep problems due to factors such as fear of death and uncertainty about anesthesia before surgery, significant decreases in sleep quality are observed after surgery due to reasons such as pain, anxiety and hospitalization. This sleeplessness can lead to many negative consequences such as delayed wound healing, increased pain, tension and difficulty in compliance with treatment. Sleep disorders also increase patients' stress and reduce their resistance. Progressive relaxation exercises (PGE) are a method that provides relaxation throughout the body by tensing and then relaxing all muscle groups in the body. This method is used as an effective nursing intervention, especially in the management of diseases and symptoms. This study aims to evaluate the effects of progressive relaxation exercises on sleep quality in patients undergoing urological surgery.

ELIGIBILITY:
Inclusion Criteria:

* • Patients must be over 18 and under 70 years old,

  * Patients must not have any visual or auditory problems that would prevent them from expressing their sleep status correctly and understanding the information provided,
  * Not have benefited from techniques such as meditation, hypnosis, yoga for up to 6 months before the study,
  * Not have a neurological or psychiatric disease,
  * Not have a sleep apnea syndrome/not have a sleep disorder diagnosis or are not receiving medical treatment for this purpose,
  * Patients must not have developed any complications within three days before, during, and after surgery,

Exclusion Criteria:

* • Those with serious cognitive disorders

  * Those with severe psychiatric disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Richard's Campbell sleep scale | 1 hour before surgery
  It was developed by Richards in 1987 and examines the previous night's sleep in 6 parameters: sleep depth, falling asleep, frequency of waking, duration of wakefulness, quality of sleep, noise level, and is scored between 100 'very appropriate' and '0' 'not appropriate'. The higher the score received from the scale, the higher the patient's sleep quality is considered.

SECONDARY OUTCOMES:
Richard's Campbell sleep scale | the night before surgery
  It was developed by Richards in 1987 and examines the previous night's sleep in 6 parameters: sleep depth, falling asleep, frequency of waking, duration of wakefulness, quality of sleep, noise level, and is scored between 100 'very appropriate' and '0' 'not appropriate'. The higher the score received from the scale, the higher the patient's sleep quality is considered.

CONTACTS AND LOCATIONS:
Overall Officials: naile akıncı, Dr., Principal Investigator — Fenerbahçe University
Locations (1):
- Atlas University, Istanbul, Turkey (Türkiye)